CLINICAL TRIAL: NCT06491420
Title: Is There a Role for Hip Arthroscopy in Patients With Femoral Head Fractures?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-038-2024
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Femur Head Fracture; Arthroscopy
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Intervention Model Description: A single limb interventional study where all cases presenting with pipkin 1 fractures are treated with arthroscopy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pipin 1 fractures fixed with arthroscopy (Experimental): Accurate portal placement was essential for optimal visualization and safe access to the hip joint.
  * The anterolateral, anterior, and distal lateral accessory portals were utilized for arthroscopic labral repair.
  * The anterolateral portal was placed approximately 1-2 cm superior to the tip of the greater trochanter and 1-2 cm anterior, at an angle of 15° to 20° relative to the floor.
  * The anterior portal was established for visualization of the posterior-superior capsule, posterior-superior labrum, posterior recess, femoral head, ligamentum teres, and other structures.
  * The distal lateral accessory portal was placed after traction was released and the operative knee was flexed to 45°.
  After reducing the fracture under arthroscopic guidance, a guidewire fixed the fracture a cannulated screw was passed over the wire to fix the fracture.
  Interventions: Other: fixation with arthroscopy

INTERVENTIONS:
Other: fixation with arthroscopy — the pipkin fracture is fixed with the help of arthroscopy and percutaneous methods.

SUMMARY:
Femoral head fractures, often caused by high-energy trauma, pose significant challenges due to complications like avascular necrosis, post-traumatic osteoarthritis, and sciatic nerve damage. While traditionally treated with open reduction and internal fixation (ORIF) or total hip replacement (THR), hip arthroscopy has emerged as a minimally invasive alternative that reduces surgical trauma, offers direct fracture visualization and manipulation, and may result in shorter recovery times and fewer complications.

DETAILED DESCRIPTION:
Femoral head fractures are uncommon but serious injuries often happen because of high-energy trauma, such as traffic accidents or falls from heights. These fractures can result in complications such as avascular necrosis (if associated with hip dislocations), post-traumatic osteoarthritis, heterotopic ossification, and sciatic nerve damage. The management of femoral head fractures is challenging and depends on several variables, such as the fracture pattern, the degree of displacement, the existence of associated injuries, and the patient's age and physical activity.

Traditionally, open reduction and internal fixation (ORIF) or total hip replacement (THR) have been the treatment of femoral head fractures, depending on the extent of the damage and the patient's expectations. However, these procedures have some drawbacks, such as increased blood loss, infection risk, surgical trauma, and implant-related complications. Furthermore, THR might not be appropriate for young, active patients who wish to maintain their natural hip joint, whereas ORIF might not be able to adequately reduce and fixate the fracture fragments, particularly in situations of comminution or impaction.

Nevertheless, hip arthroscopy has surfaced as a minimally invasive alternative for the treatment of selected femoral head fractures. Arthroscopy could be useful in femoral head fractures as it minimizes surgical aggression, in contrast to surgical hip dislocation applied in ORIF, allowing for direct control of fracture reduction, minimizing surgical morbidity, and optimizing early recovery. Hip arthroscopy allows for direct visualization and manipulation of the fracture fragments, as well as the removal of loose bodies and debris from the joint. Hip arthroscopy can also be combined with percutaneous fixation techniques to stabilize the fracture and restore joint congruence. When compared to open surgery, hip arthroscopy may offer several benefits, including shorter recovery times, less discomfort, less blood loss, and better cosmetic results. Arthroscopic-assisted percutaneous fixation has been reported as an effective treatment in selected cases of femoral head fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pipkin 1 fractures

Exclusion Criteria:

* any associated pelvic fractures
* severe medical conditions that prevent the patient from undergoing surgery
* delayed presentation after 2 weeks from initial fracture date

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Non Arthritic Hip Score | 6 months
  The Following five questions concern the amount of pain: 1 Walking on a flat surface? 2 Going up or down stairs? 3 At night while in bed? 4 Sitting or lying? 5 tanding upright? the scoring for each question is from 0 to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy-Cairo University- Faculty of Medicine, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The author will share it upon reasonable request